CLINICAL TRIAL: NCT03284437
Title: Pilot Study of Early Cognitive Training in the Intensive Care Unit
Acronym: ECTICU
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistical difficulties with implementing study.
Sponsor: Mount Carmel Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 170214-3
Record Dates: First submitted 2017-09-14; First posted 2017-09-15 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2021-07

CONDITIONS: Intensive Care Units, Delirium, Cognitive Dysfunction
MeSH Terms: conditions — Delirium; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor is not participating in patient enrollment or administration of study intervention and will not be aware of study group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (No Intervention): Usual medical care provided to patients in the ICU.
- Early Cognitive Training (Experimental): Usual medical care provided to patients in the ICU plus additional activities designed to engage the patient's attention and cognition. Activities are chosen by the family member from an activity cart according to the level designated by occupation therapy.
  Interventions: Behavioral: Early Cognitive Training

INTERVENTIONS:
Behavioral: Early Cognitive Training — Choose level of activity (e.g., coloring, holding objects) based on occupational therapist assessment.
  Arms: Early Cognitive Training

SUMMARY:
The purpose of this study is to see how early cognitive training (participation/involvement in activities to stimulate the brain) in the Intensive Care Unit (ICU) affects the number of patients who experience delirium (confusion) and cognitive impairment (problems with thinking). Reports have shown that 30% to 80% of all ICU patients will have some type of cognitive impairment: remembering, paying attention, solving problems, organizing, and working on complex tasks for some time after they leave the hospital.

Occupational therapy will do an assessment after an order is received from the doctor. The patient will be randomly placed into one of two groups. If the patient is in group A then they will continue with occupational therapy as normal. If the patient is assigned to group B then they and the family will have access to an activity cart found there in the ICU unit, directed by the nurses. The family will work with the patient on a daily basis to complete activities that are appropriate for the patient based on the occupational therapist's assessment. All patients in the study will receive medical care as usual.

Information about the patient's recovery in the hospital will be collected. In addition, patients and/or their family member will complete surveys at 6 months and 1 year after enrollment to see how they have recovered and if there are continuing issues. The two groups of patients, those who received the early cognitive training and those who did not, will be compared statistically to see if there are any differences in how well they recovered. Since this intervention involving family members working with the patient has not previously been evaluated, the study will also examine the feasibility of conducting these activities in the ICU setting.

DETAILED DESCRIPTION:
This pilot study will assess the feasibility of implementing a randomized clinical trial testing an early cognitive training program for patients in the ICU. This cognitive training program was developed at Mount Carmel Health System in conjunction with occupational therapists and has not been previously evaluated.

Specific Aim 1: To evaluate whether the trial can accrue a sufficient number of patients within a reasonable time period to complete a randomized trial for efficacy.

Specific Aim 2: To evaluate whether the trial can be conducted as designed.

Specific Aim 3: To evaluate the likelihood that the trial can retain a sufficient number of patients through the end of follow-up.

Assessments include the Montreal Cognitive Assessment Test (MoCA), Richmond Agitation and Sedation Scale (RASS), Confusion Assessment Method in the ICU (CAM-ICU) and a validated quality of life survey.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be in the intensive care unit, i.e., either the surgical intensive care unit (SICU) or medical intensive care unit (MICU).
* Patient must be ≥18 years old.
* Predicted ICU length of stay greater than 3 days.
* Patient with a RASS goal of -1 to +1 at time of enrollment.
* Patient's family member(s) agree to do the cognitive training for a least one hour a day (a series of items meant to focus and stretch cognitive ability) while in the ICU. The hour can be done incrementally if needed. Family member should be ≥18 years old.
* Family who can return to the hospital at the 6 month mark to take a final MOCA test and complete a survey.

Exclusion Criteria:

* Patient presently on Versed, Diprivan or Ativan drips.
* Patient with a history of cognitive impairment, current psychiatric diagnosis and not stable on treatment, or developmental delay.
* Patient with Alzheimer's or dementia.
* Patient with known active substance abuse.
* Patients without family support.
* Patients without the ability to return to the hospital for the 6 month visit.
* Patient with history of critical care illness within the last year from time of enrollment.
* Patients who have been critically ill for greater than 72 hours.
* Non-English speaking individuals restricting ability to follow instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Percent Enrollment | 3 Days
  Percent of eligible patients who are consented and enrolled into the study.
Percent Receiving Intervention | One month
  Percent of patients randomized to intervention who receive intervention

SECONDARY OUTCOMES:
Montreal Cognitive Assessment Score | 6 months
  Change in Montreal Cognitive Assessment score from baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Terri Swan, BSN, Principal Investigator — Mount Carmel Health System

IPD SHARING:
Plan to Share IPD: No
No plans to share at this time. This intervention is being evaluated for feasibility.